CLINICAL TRIAL: NCT03987451
Title: Investigation of Efficacy and Safety of Semaglutide s.c. Once-weekly Versus Placebo in Subjects With Non-alcoholic Steatohepatitis and Compensated Liver Cirrhosis
Brief Title: A Research Study on How Semaglutide Works in People With Fatty Liver Disease and Liver Damage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9931-4492; U1111-1224-4062 (Other: World Health Organization (WHO)); 2018-004484-31 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Results first posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): Dose escalation to 2.4 mg of semaglutide once-weekly
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Semaglutide placebo once-weekly
  Interventions: Drug: Placebo (semaglutide)

INTERVENTIONS:
Drug: Semaglutide — Semaglutide given subcutaneously (s.c., under the skin) once-weekly for 48 weeks
  Arms: Semaglutide
Drug: Placebo (semaglutide) — Semaglutide placebo s.c. given once-weekly for 48 weeks
  Arms: Placebo

SUMMARY:
Semaglutide is a medicine studied in patients with non-alcoholic steatohepatitis (NASH), as it may improve liver damage. Participants will either get semaglutide or placebo (a dummy medicine) - which treatment participants get is decided by chance. The study will last for about 61 weeks in total. Participants will have 10 clinic visits and 3 phone calls with the study doctor or staff during the study. Some of the clinic visits may be spread over more days. Participants will need to inject themselves with medicine under the skin. Participants will have to do this once a week for 48 weeks. The study includes magnetic resonance imaging (MRI) scans of the liver, 1 or 2 liver tissue samples, ultrasound scans of the stomach and a possible examination of the food pipe. For some tests participants may need to remove some items of clothing. Participants will stop in the study if the doctor thinks that there are any risks for their health. The information collected from participants during the study may help them and other patients with NASH in the future. Women cannot take part if pregnant, breast-feeding or planning to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-75 years (both inclusive) at the time of signing informed consent.
* Histologic evidence of NASH and fibrosis stage 4 according to the NASH CRN classification based on central pathologist evaluation of a liver biopsy obtained within 360 days prior to screening. In subjects who have never had a liver biopsy showing NASH and F4, liver stiffness above 14 kPa by FibroScan® at screening must be documented before subjects can have a trial-related liver biopsy
* A histological NAFLD activity score (NAS) equal to or above 3 with a score of 1 or more in lobular inflammation and hepatocyte ballooning based on central pathologist evaluation
* Body mass index equal to or above 27 kg/m^2

Exclusion Criteria:

* Presence or history of hepatic decompensation (e.g. ascites, variceal bleeding, hepatic encephalopathy or spontaneous bacterial peritonitis) or liver transplantation
* Presence or history of gastroesophageal varices within the past 360 days prior to screening. For subjects with no known history of gastroesophageal varices and with a Fibroscan® equal to or above 20 kPa and thrombocytes equal to or below 150,000, a esophagogastroduodenoscopy must be performed to evaluate presence of gastroesophageal varices
* Presence or history of hepatocellular carcinoma
* Treatment with vitamin E (at doses equal to or above 800 IU/day) or pioglitazone which has not been at a stable dose in the opinion of the investigator in the period from 90 days prior to screening
* Treatment with glucagon-like peptide-1 receptor agonists (GLP-1 RAs) in the period from 90 days prior to screening
* Treatment with other glucose lowering agent(s) (apart from what is listed in the exclusion criterion above) or weight loss medication not stable in the opinion of the investigator in the period from 28 days prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (38):
- United States (24):
  - Arizona Liver Health, Chandler, Arizona
  - The Institute for Liver Health dba Arizona Liver Health, Peoria, Arizona
  - Southern California Research Center, Coronado, California
  - Altman Clinical Translational Research Institute, La Jolla, California
  - Inland Empire Clinical Trials LLC, Rialto, California
  - Excel Medical Center Clinical Trials, LLC, Boca Raton, Florida
  - University of Florida-CTRB, Gainesville, Florida
  - University of Miami/Schiff Center for Liver Diseases, Miami, Florida
  - Piedmont Research Institute, Atlanta, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Digestive Research Alliance of Michiana, South Bend, Indiana
  - University of Kentucky Hospital, Lexington, Kentucky
  - Mercy Medical Center, GI Research, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Duke University, Durham, North Carolina
  - Gastroenterology Center For The Mid-South, Germantown, Tennessee
  - Digestive Health Research - Tristar Summit Medical Center, Hermitage, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - The University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
  - VCU Health Systems, Richmond, Virginia
- France (5):
  - Hôpital Beaujon, Clichy
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Cochin, Paris
  - Groupe Hospitalier PITIE-SALPETRIERE, Paris
  - Groupe Hospitalier Mutualiste des Portes du Sud, Vénissieux
- Germany (3):
  - Hepatologie Universitätsklinikum Frankfurt/M, Frankfurt
  - Universitätsklinikum Leipzig, Klinik und Poliklinik, Leipzig
  - Universitätsmedizin der Johannes-Gutenberg-Universität Mainz, Mainz
- Spain (2):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Virgen del Rocío, Seville
- United Kingdom (4):
  - New Queen Elizabeth Hospital Birmingham, Birmingham
  - Liver Research, London
  - Freeman Hospital, Newcastle, Newcastle upon Tyne
  - Nottingham University Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Background] Loomba R, Abdelmalek MF, Armstrong MJ, Jara M, Kjaer MS, Krarup N, Lawitz E, Ratziu V, Sanyal AJ, Schattenberg JM, Newsome PN; NN9931-4492 investigators. Semaglutide 2.4 mg once weekly in patients with non-alcoholic steatohepatitis-related cirrhosis: a randomised, placebo-controlled phase 2 trial. Lancet Gastroenterol Hepatol. 2023 Jun;8(6):511-522. doi: 10.1016/S2468-1253(23)00068-7. Epub 2023 Mar 16. PMID 36934740

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 38 sites in 5 countries as follows (number of sites that screened subjects/ number of sites that randomised subjects): United States (24/19); United Kingdom (4/3); Germany (3/2); France (5/3); Spain (2/2).
Pre-assignment Details: Participants were randomised in a 2:1 ratio to receive once-weekly either semaglutide or placebo subcutaneously as an adjunct to a reduced-calorie diet and increased physical activity.
Groups:
- Semaglutide 2.4 mg: Participants were to receive once weekly subcutaneous (s.c.) injection of semaglutide for 48 weeks. Participants initially received 0.24 milligrams (mg) of semaglutide and the dose was then escalated once in 4 weeks until the target dose of 2.4 mg was reached: 0.24 mg (week 1 to week 4), 0.5 mg (week 5 to week 8), 1.0 mg (week 9 to week 12), 1.7 mg (week 13 to week 16), 2.4 mg (week 16 to week 48).
- Placebo: Participants were to receive once weekly s.c. injection of placebo matched to semaglutide (0.24 mg, 0.5 mg, 1.0 mg, 1.7 mg or 2.4 mg) for 48 weeks.
Period: Overall Study
Arm/Group | Semaglutide 2.4 mg | Placebo
Started | 47 | 24
Completed | 45 | 23
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide 2.4 mg | Placebo | Total
Number analyzed (Participants) | 47 | 24 | 71
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 37 | 18 | 55
  65<= to <75 years | 10 | 6 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 18 | 49
  Male | 16 | 6 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 4 | 15
  Not Hispanic or Latino | 33 | 19 | 52
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 41 | 21 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With At Least One Stage of Liver Fibrosis Improvement With No Worsening of Non-Alcoholic Steatohepatitis (NASH) After 48 Weeks
Description: NASH resolution defined by NASH clinical research network (CRN) as lobular inflammation of 0 or 1; hepatocellular ballooning reduced to 0; both criteria were necessary conditions. Hepatocellular ballooning ranges from 0-2; lobular inflammation ranges from 0-3, higher scores indicating more severe hepatocellular ballooning/lobular inflammation. Worsening of NASH defined by NASH CRN as increase of at least 1 stage of either lobular inflammation, hepatocyte ballooning or steatosis. Worsening of fibrosis defined by increase in fibrosis at least 1 stage of Kleiner fibrosis classification: fibrosis stages range from 0-4, higher scores indicating greater fibrosis (0=None, 4=Cirrhosis). Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Week 48
Population: Full analysis set (FAS) included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 47 | 24
Percentage of participants | 10.6 | 29.2
Statistical Analysis 1: Comparison: Semaglutide 2.4 mg vs Placebo; The common odds ratio between semaglutide and placebo adjusting for baseline diabetes was estimated along with exact 95% confidence interval based on conditioning on the marginal 2×2 tables; Test type: Superiority; p = 0.0867, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.28, 95% CI 2-sided [0.06 to 1.24]

2. Secondary Outcome: Change From Baseline in Liver Fat Content Measured by Magnetic Resonance Imaging-Proton Density Fat Fraction (MRI-PDFF)-Ratio to Baseline
Description: Change in liver fat content (measured as percentage) from baseline to week 48 is presented as ratio to baseline. Liver fat content was assessed via MRI-PDFF technique and results were measured in percentage. MRI-PDFF utilized a gradient echo sequence with low flip angle to minimize T1 bias, corrected T2* decay (due to iron overload) via modeling of the fat signal as a superposition of multiple frequency components from 5 different lipid types, and was applied in each of the 9 Couinaud segments. This technique improved fat quantification accuracy for the entire liver permitting quantification of small differences/changes following pharmacological intervention. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: FAS included all randomised participants. Overall number of participants analysed = Number of participants who contributed to the analysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of liver fat content
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 38 | 18
Ratio of liver fat content | 0.62 (63.38) | 1.01 (34.46)

3. Secondary Outcome: Change From Baseline in Liver Stiffness Measured by Magnetic Resonance Elastography (MRE)-Ratio to Baseline
Description: Change in Liver Stiffness from baseline to week 48 is presented as ratio to baseline. Liver stiffness was measured in kilopascal using MRE. MRE is a technology that uses MRI imaging with low-frequency vibrations to create a visual map (elastogram) that shows stiffness of the liver. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of liver stiffness
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 35 | 21
Ratio of liver stiffness | 0.87 (22.24) | 0.98 (28.51)

4. Secondary Outcome: Percentage of Participants With NASH Resolution After 48 Weeks
Description: NASH resolution defined by NASH clinical research network as lobular inflammation of 0 or 1 and hepatocellular ballooning reduced to 0; both criteria were necessary conditions. Hepatocellular ballooning ranges from 0-2; lobular inflammation ranges from 0-3, with higher scores indicating more severe hepatocellular ballooning or lobular inflammation. Worsening of fibrosis defined by an increase in fibrosis at least one stage of Kleiner fibrosis classification: fibrosis stages range from 0-4, with higher scores indicating greater fibrosis (0=None, 4=Cirrhosis). Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Week 48
Population: FAS included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 47 | 24
Percentage of participants | 34.0 | 20.8

5. Secondary Outcome: Change From Baseline in Fibrosis-4 Score-Ratio to Baseline
Description: Change in fibrosis-4 score from baseline to week 48 is presented as ratio to baseline. Fibrosis-4 is the ratio of age in years and aminotransferase to platelet count. It is a non-invasive hepatic fibrosis index score combining standard biochemical values, platelets, alanine aminotransferase (ALT), aspartate aminotransferase (AST) and age that was calculated using formula: Fibrosis-4 = (Age [years] x AST [units per liter (U/L)]) / (platelets [10^9 cells/L] x (square root of ALT [U/L])). A Fibrosis-4 index of < 1.45 indicated no or moderate fibrosis and an index of > 3.25 indicated extensive fibrosis/cirrhosis. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fibrosis-4 score
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 44 | 23
Ratio of fibrosis-4 score | 0.9 (30.7) | 1.0 (38.0)

6. Secondary Outcome: Percentage of Participants With Change in Non-Alcoholic Fatty Liver Disease (NAFLD) Activity Score (NAS)
Description: Percentage of participants who had worsened, improved or had no change in total NAS from baseline to week 48 or missing data is presented. Worsening was defined as an increase of at least 1 in the NAS; Improvement was defined as a decrease of at least 1 in the NAS; while no change corresponds to no change in NAS and missing refers to participants with missing outcomes for NAS from baseline to week 48. NAS was calculated as the sum of scores for steatosis (0 to 3), lobular inflammation (0 to 3), and hepatocyte ballooning (0 to 2). Therefore, it is assessed on a scale of 0-8, with higher scores indicating more severe disease. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: FAS included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 47 | 24
Percentage of participants
  Improvement | 61.7 | 58.3
  Worsening | 2.1 | 16.7
  No change | 21.3 | 20.8
  Missing | 14.9 | 4.2

7. Secondary Outcome: Percentage of Participants With Change in The Fibrosis Stage According to The Kleiner Fibrosis Classification
Description: Percentage of participants who had improved, worsened, or had no change in fibrosis stage from baseline to week 48 or missing data is presented. The degree of fibrosis was described by the Kleiner fibrosis staging system, ranging from F0 (absence of fibrosis), F1 (portal/perisinusoidal fibrosis), F2 (perisinusoidal and portal/periportal fibrosis), F3 (septal or bridging fibrosis) through F4 (cirrhosis). Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: FAS included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 47 | 24
Percentage of participants
  Improvement | 12.8 | 33.3
  Worsening | 0.0 | 0.0
  No change | 72.3 | 62.5
  Missing | 14.9 | 4.2

8. Secondary Outcome: Percentage of Participants With Change in Hepatocyte Ballooning
Description: Percentage of participants who had improved, worsened, or had no change in hepatocyte ballooning from baseline to week 48 or missing data is presented. Hepatocyte ballooning was assessed on a scale of 0-2, with higher scores indicating more severe disease. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: FAS included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 47 | 24
Percentage of participants
  Improvement | 55.3 | 33.3
  Worsening | 2.1 | 8.3
  No change | 27.7 | 54.2
  Missing | 14.9 | 4.2

9. Secondary Outcome: Percentage of Participants With Change in Lobular Inflammation
Description: Percentage of participants who had improved, worsened, or had no change in lobular inflammation from baseline to week 48 or missing data is presented. Lobular inflammation was assessed on a scale of 0-3, with higher scores indicating more severe lobular inflammation. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: FAS included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 47 | 24
Percentage of participants
  Improvement | 42.6 | 37.5
  Worsening | 12.8 | 12.5
  No change | 29.8 | 45.8
  Missing | 14.9 | 4.2

10. Secondary Outcome: Percentage of Participants With Change in Steatosis
Description: Percentage of participants who had improved, worsened, or had no change in steatosis from baseline to week 48 or missing data is presented. Steatosis was assessed on a scale of 0-3, with higher scores indicating more severe steatosis. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: FAS included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 47 | 24
Percentage of participants
  Improvement | 44.7 | 33.3
  Worsening | 2.1 | 16.7
  No change | 38.3 | 45.8
  Missing | 14.9 | 4.2

11. Secondary Outcome: Percentage of Participants With Change in The Steatosis-Activity-Fibrosis (SAF) Activity Component Score
Description: Percentage of participants who had improved, worsened, or had no change in the activity component of the SAF score from baseline to week 48 or missing data is presented. SAF score was assessed on a scale of 0-4, with higher scores indicating more severe disease. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: FAS included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 47 | 24
Percentage of participants
  Improvement | 57.4 | 50.0
  Worsening | 8.5 | 12.5
  No change | 19.1 | 33.3
  Missing | 14.9 | 4.2

12. Secondary Outcome: Percentage of Participants With Change in The Ishak Fibrosis Score
Description: Percentage of participants who had improved, worsened, or had no change in the Ishak fibrosis score from baseline to week 48 or missing data is presented. Ishak fibrosis score was assessed on a scale of 0-6, with higher scores indicating more severe disease. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: FAS included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 47 | 24
Percentage of participants
  Improvement | 27.7 | 37.5
  Worsening | 2.1 | 12.5
  No change | 55.3 | 45.8
  Missing | 14.9 | 4.2

13. Secondary Outcome: Change From Baseline in Hepatic Collagen
Description: Change in hepatic collagen from baseline to week 48 was analysed. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of hepatic collagen
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 37 | 21
Percentage of hepatic collagen | -1.7 (7.9) | -1.2 (5.1)

14. Secondary Outcome: Percentage of Participants With Improvement in Fibrosis Stage According to The Kleiner Fibrosis Classification (Yes/No)
Description: Improvement is defined as at least one stage decrease from baseline to week 48 in Kleiner fibrosis classification. The degree of fibrosis was described by the Kleiner fibrosis staging system, ranging from F0 (absence of fibrosis), F1 (portal/perisinusoidal fibrosis), F2 (perisinusoidal and portal/periportal fibrosis), F3 (septal or bridging fibrosis) through F4 (cirrhosis). Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: FAS included all randomised participants. In below table, 'Yes' infers percentage of participants who achieved at least one stage decrease from baseline to week 48 in Kleiner fibrosis classification; 'No' infers vice-versa; 'Missing' refers to percentage of participants with data missing due to different reasons (lost to follow-up, withdrawal).
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 47 | 24
Percentage of participants
  Yes | 12.8 | 33.3
  No | 72.3 | 62.5
  Missing | 14.9 | 4.2

15. Secondary Outcome: Percentage of Participants With Improvement in Hepatocyte Ballooning (Yes/No)
Description: Improvement is defined as at least one stage decrease from baseline to week 48 in hepatocyte ballooning clinical research network (CRN) score. Hepatocyte ballooning was assessed on a scale of 0-2, with higher scores indicating more severe disease. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: FAS included all randomised participants. In below table, 'Yes' infers percentage of participants who achieved at least one stage decrease from baseline to week 48 in hepatocyte ballooning; 'No' infers vice-versa; 'Missing' refers to percentage of participants with data missing due to different reasons (lost to follow-up, withdrawal).
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 47 | 24
Percentage of participants
  Yes | 55.3 | 33.3
  No | 29.8 | 62.5
  Missing | 14.9 | 4.2

16. Secondary Outcome: Percentage of Participants With Improvement in Lobular Inflammation (Yes/No)
Description: Improvement is defined as at least one stage decrease from baseline to week 48 in lobular inflammation CRN score. Lobular inflammation was assessed on a scale of 0-3, with higher scores indicating more severe lobular inflammation. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: FAS included all randomised participants. In below table, 'Yes' infers percentage of participants who achieved at least one stage decrease from baseline to week 48 in lobular inflammation; 'No' infers vice-versa; 'Missing' refers to percentage of participants with data missing due to different reasons (lost to follow-up, withdrawal).
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 47 | 24
Percentage of participants
  Yes | 42.6 | 37.5
  No | 42.6 | 58.3
  Missing | 14.9 | 4.2

17. Secondary Outcome: Percentage of Participants With Improvement in Steatosis (Yes/No)
Description: Improvement is defined as at least one stage decrease from baseline to week 48 in steatosis CRN score. Steatosis was assessed on a scale of 0-3, with higher scores indicating more severe steatosis. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: FAS included all randomised participants. In below table, 'Yes' infers percentage of participants who achieved at least one stage decrease from baseline to week 48 in steatosis; 'No' infers vice-versa; 'Missing' refers to percentage of participants with data missing due to different reasons (lost to follow-up, withdrawal).
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 47 | 24
Percentage of participants
  Yes | 44.7 | 33.3
  No | 40.4 | 62.5
  Missing | 14.9 | 4.2

18. Secondary Outcome: Percentage of Participants With Improvement in NAS (Yes/No)
Description: Improvement is defined as at least one stage decrease from baseline to week 48 in NAS. NAS was calculated as the sum of scores for steatosis (0 to 3), lobular inflammation (0 to 3), and hepatocyte ballooning (0 to 2). Therefore, it is assessed on a scale of 0-8, with higher scores indicating more severe disease. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: FAS included all randomised participants. In below table, 'Yes' infers percentage of participants who achieved at least one stage decrease from baseline to week 48 in NAS; 'No' infers vice-versa; 'Missing' refers to percentage of participants with data missing due to different reasons (lost to follow-up, withdrawal).
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 47 | 24
Percentage of participants
  Yes | 61.7 | 58.3
  No | 23.4 | 37.5
  Missing | 14.9 | 4.2

19. Secondary Outcome: Percentage of Participants With Improvement in SAF Activity Component Score (Yes/No)
Description: Improvement is defined as at least one stage decrease from baseline to week 48 in SAF score. SAF score was assessed on a scale of 0-4, with higher scores indicating more severe disease. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: FAS included all randomised participants. In below table, 'Yes' infers percentage of participants who achieved at least one stage decrease from baseline to week 48 in SAF score; 'No' infers vice-versa; 'Missing' refers to percentage of participants with data missing due to different reasons (lost to follow-up, withdrawal).
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 47 | 24
Percentage of participants
  Yes | 57.4 | 50.0
  No | 27.7 | 45.8
  Missing | 14.9 | 4.2

20. Secondary Outcome: Percentage of Participants With Improvement in Ishak Fibrosis Score (Yes/No)
Description: Improvement is defined as at least one stage decrease from baseline to week 48 in Ishak fibrosis score. Ishak fibrosis score was assessed on a scale of 0-6, with higher scores indicating more severe disease. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: FAS included all randomised participants. In below table, 'Yes' infers percentage of participants who achieved at least one stage decrease from baseline to week 48 in Ishak fibrosis score; 'No' infers vice-versa; 'Missing' refers to percentage of participants with data missing due to different reasons (lost to follow-up, withdrawal).
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 47 | 24
Percentage of participants
  Yes | 27.7 | 37.5
  No | 57.4 | 58.3
  Missing | 14.9 | 4.2

21. Secondary Outcome: Change From Baseline in Body Weight
Description: Change in body weight from baseline to week 48 is presented. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 46 | 23
Kilograms | -8.6 (7.8) | -0.8 (5.0)

22. Secondary Outcome: Relative Change From Baseline in Body Weight
Description: Relative change in body weight (measured as kg) from baseline to week 48 is presented. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: FAS included all randomised participants.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 47 | 24
percent change | -8.83 (7.44) | -0.09 (7.44)

23. Secondary Outcome: Change From Baseline in Waist Circumference
Description: Change in waist circumference from baseline to week 48 is presented. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 45 | 22
centimeters | -6.3 (7.7) | 0.4 (6.8)

24. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: Change in BMI from baseline to week 48 is presented. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilograms per meter square
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 46 | 23
Kilograms per meter square | -3.1 (2.8) | -0.2 (1.8)

25. Secondary Outcome: Percentage of Participants With Weight Loss of >= 5% of Baseline Body Weight at Week 48
Description: Percentage of participants with weight loss of greater than or equal to (≥) 5% of baseline body weight at 48 weeks is presented. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Week 48
Population: FAS included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 47 | 24
Percentage of participants | 62.0 | 25.4

26. Secondary Outcome: Percentage of Participants With Weight Loss of >= 10% of Baseline Body Weight at Week 48
Description: Percentage of participants with weight loss of ≥ 10% of baseline body weight at 48 weeks is presented. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Week 48
Population: FAS included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 47 | 24
Percentage of participants | 40.5 | 0

27. Secondary Outcome: Change From Baseline in Glycosylated Haemoglobin A1c (HbA1c)
Description: Change in HbA1c from baseline to week 48 is presented. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: FAS included all randomised participants. Overall number of participants analysed = Number of participants with type 2 diabetes who contributed to the analysis
Measure: Mean (Standard Deviation); unit: Percentage of HbA1C
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 34 | 18
Percentage of HbA1C | -1.4 (1.1) | 0.2 (1.1)

28. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Change in FPG from baseline to week 48 is presented. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 31 | 16
millimoles per liter (mmol/L) | -2.20 (2.52) | 0.23 (2.94)

29. Secondary Outcome: Change From Baseline in Fasting C-peptide-Ratio to Baseline
Description: Change in fasting C-peptide [measured as nanomoles per litre (nmol/L)] from baseline to week 48 is presented as ratio to baseline. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting C-peptide
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 31 | 16
Ratio of fasting C-peptide | 0.95 (47.08) | 1.00 (45.73)

30. Secondary Outcome: Change From Baseline in Systolic And Diastolic Blood Pressure
Description: Change in systolic and diastolic blood pressure from baseline to week 48 is presented. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeter of mercury
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 46 | 23
millimeter of mercury
  Change From Baseline in Systolic Blood Pressure | -4.1 (17.6) | 0.1 (17.1)
  Change From Baseline in Diastolic Blood Pressure | 0.4 (11.7) | -0.7 (8.4)

31. Secondary Outcome: Change From Baseline in Total Cholesterol-Ratio to Baseline
Description: Change in total cholesterol (measured as mmol/L) from baseline to week 48 is presented as ratio to baseline. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 44 | 21
Ratio of total cholesterol | 0.98 (11.86) | 1.05 (17.61)

32. Secondary Outcome: Change From Baseline in Low-Density Lipoprotein (LDL) Cholesterol-Ratio to Baseline
Description: Change in LDL cholesterol (measured as mmol/L) from baseline to week 48 is presented as ratio to baseline. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 44 | 21
Ratio of LDL cholesterol | 0.99 (17.88) | 1.02 (30.07)

33. Secondary Outcome: Change From Baseline in High-Density Lipoprotein (HDL) Cholesterol-Ratio to Baseline
Description: Change in HDL cholesterol (measured as mmol/L) from baseline to week 48 is presented as ratio to baseline. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 44 | 21
Ratio of HDL cholesterol | 1.07 (12.83) | 0.99 (16.30)

34. Secondary Outcome: Change From Baseline in Very Low-Density Lipoprotein (VLDL) Cholesterol-Ratio to Baseline
Description: Change in VLDL cholesterol (measured as mmol/L) from baseline to week 48 is presented as ratio to baseline. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of VLDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 44 | 21
Ratio of VLDL cholesterol | 0.90 (28.37) | 1.09 (28.09)

35. Secondary Outcome: Change From Baseline in Triglycerides-Ratio to Baseline
Description: Change in triglycerides (measured as mmol/L) from baseline to week 48 is presented as ratio to baseline. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 44 | 21
Ratio of triglycerides | 0.90 (28.40) | 1.09 (28.08)

36. Secondary Outcome: Change From Baseline in Free Fatty Acids (FFA)-Ratio to Baseline
Description: Change in free fatty acids (measured as mmol/L) from baseline to week 48 is presented as ratio to baseline. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of FFA
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 42 | 21
Ratio of FFA | 1.07 (75.99) | 1.43 (77.70)

37. Secondary Outcome: Change From Baseline in High-Sensitivity C-reactive Protein (hsCRP)-Ratio to Baseline
Description: Change in hsCRP (measured as milligrams per liter) from baseline to week 48 is presented as ratio to baseline. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of hsCRP
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 46 | 23
Ratio of hsCRP | 0.63 (107.66) | 1.13 (70.38)

38. Secondary Outcome: Change From Baseline in Alanine Aminotransferase (ALT)-Ratio to Baseline
Description: Change in ALT (measured as units per liter) from baseline to week 48 is presented as ratio to baseline. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of ALT
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 46 | 23
Ratio of ALT | 0.7 (58.1) | 1.0 (32.2)

39. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase (AST)-Ratio to Baseline
Description: Change in AST (measured as units per liter) from baseline to week 48 is presented as ratio to baseline. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AST
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 46 | 23
Ratio of AST | 0.7 (47.8) | 1.0 (29.0)

40. Secondary Outcome: Change From Baseline in Gamma-Glutamyl Transferase (GGT)-Ratio to Baseline
Description: Change in GGT (measured as units per liter) from baseline to week 48 is presented as ratio to baseline. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of GGT
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 46 | 23
Ratio of GGT | 0.7 (40.9) | 1.0 (24.4)

41. Secondary Outcome: Change From Baseline in Albumin-Ratio to Baseline
Description: Change in albumin [measured as grams per deciliter (g/dL)] from baseline to week 48 is presented as ratio to baseline. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of albumin
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 46 | 23
Ratio of albumin | 1.0 (6.1) | 1.0 (5.9)

42. Secondary Outcome: Changes From Baseline in Thrombocytes-Ratio to Baseline
Description: Change in thrombocytes [measured as 10^9 cells per liter] from baseline to week 48 is presented as ratio to baseline. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of thrombocytes
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 46 | 23
Ratio of thrombocytes | 1.0 (16.1) | 1.0 (14.7)

43. Secondary Outcome: Change From Baseline in International Normalized Ratio (INR)-Ratio to Baseline
Description: Change in INR from baseline to week 48 is presented as ratio to baseline. INR is the ratio of measured prothrombin time over normal prothrombin time and it evaluates the extrinsic coagulation pathway (vitamin K dependent clotting factors II; V, VII, IX and X). These clotting factors are synthesised in the liver, thus INR is used as a marker of liver synthesis function. The therapeutic INR range varies, most commonly an INR 2-3 goal, but ranging from 1.5-4.0. Bleeding complications are more likely to occur above an INR value of 4.0. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of INR
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 46 | 22
Ratio of INR | 1.02 (5.59) | 1.01 (25.07)

44. Secondary Outcome: Change From Baseline in Direct Bilirubin-Ratio to Baseline
Description: Change in direct bilirubin [measured as micromoles per liter (umol/L)] from baseline to week 48 is presented as ratio to baseline. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of direct bilirubin
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 45 | 22
Ratio of direct bilirubin | 1.1 (33.7) | 1.0 (24.8)

45. Secondary Outcome: Change From Baseline in Total Bilirubin-Ratio to Baseline
Description: Change in total bilirubin [measured as umol/L] from baseline to week 48 is presented as ratio to baseline. Outcome measure was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (week 55); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 48
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total bilirubin
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 46 | 23
Ratio of total bilirubin | 1.0 (34.5) | 0.9 (24.5)

46. Secondary Outcome: Number of Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical trial participant administered or using a medicinal product, whether or not considered related to the medicinal product or usage. All AEs reported here are TEAEs. TEAE is defined as an event that had onset date during the on-treatment period. Outcome measure was evaluated based on data from on-treatment period which started on the date of first administration of trial product and ended on the date of whatever comes first of: a) last dose of trial product + 49 days (7 half-lives of semaglutide), b) follow-up visit (week 55), or c) end of the in-trial period.
Time Frame: From baseline (week 0) to week 55
Population: Safety analysis set included all participants that received at least one dose of randomised treatment.
Measure: Number; unit: Events
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 47 | 24
Events | 290 | 85

47. Secondary Outcome: Number of Treatment-Emergent Hypoglycaemic Episodes
Description: Hypoglycaemic episode (blood glucose less than or equal to (<=) 3.9 mmol/L [70 milligrams per decilitre (mg/dL)] Or greater than (>) 3.9 mmol/L (70 mg/dL) occurring in conjunction with hypoglycaemic symptoms) is defined as treatment emergent if the onset of the episode occurs during the on-treatment period. Outcome measure was evaluated based on data from on-treatment period which started on the date of first administration of trial product and ended on the date of whatever comes first of: a) last dose of trial product + 49 days (7 half-lives of semaglutide), b) follow-up visit (week 55), or c) end of the in-trial period.
Time Frame: From baseline (week 0) to week 55
Population: Safety analysis set included all participants that received at least one dose of randomised treatment. Overall number of participants analysed = Number of participants with type 2 diabetes who contributed to the analysis
Measure: Number; unit: Episodes
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 35 | 18
Episodes | 34 | 15

48. Secondary Outcome: Change From Baseline in Pulse
Description: Change in pulse from baseline to week 48 is presented. Outcome measure was evaluated based on data from on-treatment period which started on the date of first administration of trial product and ended on the date of whatever comes first of: a) last dose of trial product + 49 days (7 half-lives of semaglutide), b) follow-up visit (week 55), or c) end of the in-trial period.
Time Frame: Baseline (week 0), Week 48
Population: Safety analysis set included all participants that received at least one dose of randomised treatment. Overall number of participants analysed = Number of participants who contributed to the analysis
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 35 | 17
Beats per minute | 6 (11) | 2 (14)

ADVERSE EVENTS:
Time Frame: From week 0 to week 55. Results are based on the safety analysis set which included all participants who received at least one dose of randomised treatment.
Description: All AEs reported here are TEAEs. TEAE is defined as an event that had onset date during on-treatment period. On-treatment period which started on the date of first administration of trial product and ended on the date of whatever comes first of: a) last dose of trial product + 49 days (7 half-lives of semaglutide), b) follow-up visit (week 55), or c) end of the in-trial period (week 55).
Arm/Group | Semaglutide 2.4 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/24
Serious Adverse Events (participants affected / at risk) | 6/47 | 2/24
Other Adverse Events (participants affected / at risk) | 38/47 | 15/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 2.4 mg (N=47) | Placebo (N=24)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal claudication (Nervous system disorders) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Vitreous detachment (Eye disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 2.4 mg (N=47) | Placebo (N=24)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 5 (8) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 9 (13) | 2 (3)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Eructation (Gastrointestinal disorders) | 6 (19) | 0 (0)
Fatigue (General disorders) | 4 (7) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 21 (34) | 4 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3) | 4 (4)
Vomiting (Gastrointestinal disorders) | 8 (10) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property

DOCUMENTS (2):
  • Study Protocol (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/51/NCT03987451/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/51/NCT03987451/SAP_001.pdf